CLINICAL TRIAL: NCT03335072
Title: Kebele Elimination of Trachoma for Ocular Health
Acronym: KETFO
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Eye Institute (NEI) (NIH); Eyu-Ethiopia (Unknown); Bahir Dar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-22201; 1UG1EY028088 (NIH)
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Trachoma
Keywords: Azithromycin; Mass Drug Administration; Antibiotic Resistance
MeSH Terms: conditions — Trachoma | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- WHO-recommended (Active Comparator): Annual mass azithromycin distribution of all residents
  Interventions: Drug: Azithromycin
- Age-based core group (Experimental): Annual mass azithromycin treatment of everyone plus quarterly treatment of children
  Interventions: Drug: Azithromycin
- PCR infection-based core group (Experimental): Annual mass azithromycin treatment plus quarterly treatment of a PCR-based cohort that would be a subset of the age-based core group.
  Interventions: Drug: Azithromycin
- TI-based core group (Experimental): Annual mass azithromycin treatment plus quarterly treatment of a conjunctival photography-based cohort that would be a subset of the age-based core group
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Mass Drug Administration
  Other Names: Zithromax

SUMMARY:
The investigators propose a cluster-randomized clinical trial to determine whether an intensive, targeted azithromycin distribution strategy is effective for elimination of trachoma at the kebele level compared to the World Health Organization (WHO) recommendation of annual azithromycin distribution.

DETAILED DESCRIPTION:
The investigators propose to randomize at the kebele level, which consist of approximately 15 villages, 4,000 residents, and are served by a single primary school. Eighty kebeles will be randomized to one of four arms: 1) annual mass azithromycin distribution per WHO guidelines (Annual); 2) annual mass azithromycin distribution plus quarterly targeted treatment of all children aged 0-9 years (Core Group-Age); 3) annual mass azithromycin distribution plus quarterly targeted treatment of all children aged 0-9 years with a positive chlamydial PCR test (Core Group-PCR); or 4) annual mass azithromycin distribution plus quarterly targeted treatment of all children aged 0-9 years positive for conjunctival inflammation as assessed from annual photography (Core Group-TI). The primary outcome for the trial will be the ocular chlamydia prevalence at 12, 24, and 36 months. Secondary outcomes will include bacterial load of ocular chlamydia via quantitative PCR, the prevalence of clinically active trachoma assessed at 12, 24, and 36 months, and serology via dried blood spot at baseline and 36 months.

ELIGIBILITY:
Inclusion Criteria:

* All individuals in all communities will be eligible for annual mass azithromycin distribution per WHO guidelines.

Exclusion Criteria:

* Those who do not consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320000 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Ocular chlamydia measured in a population based age-stratified sample of the entire community | 36 months
  Assessed by PCR

SECONDARY OUTCOMES:
Infectious load of chlamydia among 0-9 year-old children infected with ocular chlamydia | 36 months
  Assessed by PCR
Conjunctival inflammation | 36 months
  Assessed from conjunctival photography

CONTACTS AND LOCATIONS:
Overall Officials: Tom M Lietman, MD, Principal Investigator — University of California, San Francisco; Hadley Burroughs, MSPH, Study Director — University of California, San Francisco
Locations (2):
- UCSF Proctor Foundation, San Francisco, California, United States
- Eyu-Ethiopia, Bahir Dar, Ethiopia

IPD SHARING:
Plan to Share IPD: No